CLINICAL TRIAL: NCT00000254
Title: Isoflurane at Subanesthetic Concentrations
Brief Title: Isoflurane at Subanesthetic Concentrations - 6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NIDA-08391-6; R01DA008391 (NIH); R01-08391-6
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: isoflurane; general anesthetic; inhalant; subjective effects; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Nitrous Oxide; Isoflurane

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- 0% isoflurane (Sham Comparator)
  Interventions: Drug: 40% Nitrous oxide; Other: Sham comparator
- 0.2% isoflurane (Active Comparator)
  Interventions: Drug: 40% Nitrous oxide; Drug: 0.2% isoflurane
- 0.4% isoflurane (Active Comparator)
  Interventions: Drug: 40% Nitrous oxide; Drug: 0.4% isoflurane
- 0.6% isoflurane (Active Comparator)
  Interventions: Drug: 40% Nitrous oxide; Drug: 0.6% isoflurane

INTERVENTIONS:
Drug: 40% Nitrous oxide — Used as pain assay positive control
Other: Sham comparator — 0% isoflurane in oxygen
  Arms: 0% isoflurane
Drug: 0.2% isoflurane
  Arms: 0.2% isoflurane
Drug: 0.4% isoflurane
  Arms: 0.4% isoflurane
Drug: 0.6% isoflurane
  Arms: 0.6% isoflurane

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. To test the hypothesis that isoflurane at subanesthetic concentrations does not reduce cold-water immersion pain in healthy volunteers.

ELIGIBILITY:
Please contact site for information.

Ages: 21 Years to 34 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 1995-01; Primary Completion 1995-09 (Actual); Study Completion 1995-09 (Actual)

PRIMARY OUTCOMES:
Pain response | Post inhalation
  Effects of inhaled isoflurane on pain from immersion of subject's arm in ice cold water. Nitrous oxide (40%) was used as a positive control to confirm sensitivity of the pain assay.

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States

REFERENCES:
- [Background] Anesthesiology, 1995, 83: A287